CLINICAL TRIAL: NCT05931848
Title: Effects of Group Based Multimodal Exercise Training Combined With Otago Home-Based Exercise Program on Physical Performance, Balance, and Social Participation in Community-Dwelling Older Women (METCOHEP Study)
Brief Title: Otago Home-Based Exercise Program in Community-Dwelling Older Women (METCOHEP Study)
Acronym: METCOHEP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study could not be completed because of the research team was seperated.
Sponsor: Istanbul Arel University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other); Istanbul Aydın University (Other); Kadikoy Municipality Social Life Center (Unknown)
Responsible Party: Principal Investigator, NAZLI GÜNGÖR, Lecturer, Department of Physiotherapy and Rehabilitation, Faculty of Health Sciences, Istanbul Arel University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: METCOHEP
Record Dates: First submitted 2023-05-20; First posted 2023-07-05 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Balance Impairment; Risk of Falling
Keywords: community-dwelling older women; Otago exercises; physical performance; balance; social participation; randomized controlled trial
MeSH Terms: interventions — Warm-Up Exercise

STUDY DESIGN:
Intervention Model Description: clinical research/randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Otago exercise group (Experimental): The treatment program, which will last for 16 weeks, 3 days a week, a total of 48 sessions will be held. The program will be held one day a week with a maximum of 8 participants per group, under the supervision of a physiotherapist, in the Kadikoy Municipality Social Life Center, in the form of group exercise training, and two days a week at the participants' homes, with the implementation of the Otago Home Exercise Program non-supervised. Participants will be informed that the program should be implemented on non-consecutive days. All warm-up and strengthening exercises will be applied in combination with breathing. While the home exercise program is being taught to the patients, information will be given about the situations where the exercise is contraindicated and should be stopped.
  Within the scope of group exercise training, it is planned to implement a structured program of approximately 45-60 minutes, including warm-up, strengthening, balance and cool-down exercises.
  Interventions: Other: Warm-up and Cool-down Program; Other: Strengthening Exercises; Other: Balance Exercises; Other: Otago Home Exercise Program
- control group (No Intervention): The control group will not be included in any exercise program, and they will be informed that they can participate in the same program after 16 weeks if they prefer. At the same time, a one-session training will be given to all participants of intervention and control groups at the Kadıköy Municipality Social Life Center, where information about the factors that increase the risk of falling and house arrangements will be provided.

INTERVENTIONS:
Other: Warm-up and Cool-down Program — Each exercise in the warm-up and cool-down protocols consisting of active movements and static stretching exercises will be performed as 1 set and 10 repetitions. Active movements will be performed for 10 seconds. The detailed protocol is shown below.
  Neck flexion/extension/lateral flexion Circles made with the head chin-tuck Backward bilateral shoulder circumduction Shoulder external rotation with hands clasped at neck Circles with wrists clasped clockwise and counterclockwise Reciprocal upper extremity flexion-extension cat-camel Trunk lateral flexion with hands clasped overhead Trunk rotation in both directions Ankle dorsi/plantar flexion with knee extension Static Stretching Exercises Neck lateral flexor stretch Posterior capsule stretching Hands clasped trunk flexion lateral Trunk lateral flexion with hands clasped Trunk rotation in both directions Knee extensor and ankle plantar flexor stretching by reaching for toes
  Arms: Otago exercise group
Other: Strengthening Exercises — The progression of the strengthening program will be achieved by gradually changing the number of repetitions, sets, resistance and the number of exercises.
  1-6 Weeks Upper extremity strengthening in unilateral PNF D2 pattern, Scapulothoracic strengthening with shoulder extension in elbow extension, Scapulothoracic strengthening with shoulder extension in elbow flexion, hip flexor strengthening, Hip abductor strengthening in knee flexion, when sit on the chair fingertip ups and downs 7-12 Weeks Added exercises Scapular adductor strengthening with shoulders in horizontal abduction position, Shoulder adductor strengthening in elbow extension with trunk lateral flexion in arms overhead position, hip abductor strengthening 13-16 Weeks Added exercises Shoulder abductor/flexor strengthening in the scapular plane, Elbow flexor strengthening, Upper extremity strengthening in unilateral PNF D2 pattern with trunk rotation, Taking a lateral step in a mini-squat position
  Arms: Otago exercise group
Other: Balance Exercises — Balance exercises will be applied following the strengthening exercises. The exercises will be gradually made more difficult. Participants will be encouraged to complete the balance exercises by standing next to the grab bar and with as little support as possible.
  1-6. Week Rising and falling on the heels Hands at waist trunk extension hip abduction 6-9. Week Hip abduction and extension without lowering the foot to the ground, respectively 5 sec stop on tiptoe 5 seconds standing on one leg 10-12. Week Abduction, extension, and flexion of the hips without lowering the foot to the ground, respectively.
  5 sec stop on tiptoe 10 sec stop on tiptoe 5 seconds standing on one leg 10 seconds standing on one leg 13-16. Week Abduction, extension, and flexion of the hips without lowering the foot to the ground, respectively.
  10 sec stop on tiptoe 15 sec stop on tiptoe 10 seconds standing on one leg 15 seconds standing on one leg
  Arms: Otago exercise group
Other: Otago Home Exercise Program — The exercises included in the Otago Home Exercise Program will be taught to the participants after the group exercise session held at the Social Life Center. At the same time, home exercise training will be supported by brochures and videos. In addition to the exercises in the program, participants will be asked to do 30 minutes of moderate-intensity walking 2 days a week. Participants will be asked to record the exercises they did during the week in the exercise diary given to them.
  Balance Exercises
  1. Knee bend (half squat)
  2. Walking backwards
  3. Walk and turn around
  4. Sideways walking
  5. Tandem stance
  6. Tandem walking
  7. Standing on one leg
  8. Walking on the heel
  9. Toe walking
  10. Tandem walking backwards
  11. Sit down
  12. Going up and down stairs Strengthening Exercises
  1. Knee extension 2. Knee flexion 3. Hip abduction 4. Ankle plantar flexion 5. Ankle dorsiflexion
  Arms: Otago exercise group

SUMMARY:
The aim of this study is to investigate the effect of group-based multimodal exercise training combined with Otago home-based exercise program on physical performance, balance and social participation in community-dwelling older women.

Hypotheses:

H0: Group-based multimodal exercise training combined with Otago home-based exercise program in community-dwelling older women has no effect on physical performance, balance and social participation.

H1: Group-based multimodal exercise training combined with Otago home-based exercise program in community-dwelling older women has positive effects on physical performance, balance and social participation.

Within the scope of the study, the exercise program will be carried out 3 days a week and for 16 weeks;

* One day a week under the supervision of a physiotherapist, in the form of group exercise training in the center
* Two days a week, the Otago Home Exercise Program will be conducted non-supervised at the participants' homes.

Within the scope of group exercise training, it is planned to implement a program of approximately 45-60 minutes, including warm-up, strengthening, balance and cool-down exercises. The control group will not be included in any exercise application, if they wish, they can be recruited in the same program after 16 weeks. In addition, all participants will be given a training in which they will be informed about the risk of falling. There will be 2 evaluations at the beginning of the study and at the end of the 16-week program. Within the scope of the study, participants' balance, walking speed, muscle strength, fear of falling, participation, life satisfaction and loneliness parameters will be evaluated.

At the end of this study, the change in balance, walking speed, muscle strength, fear of falling, participation, life satisfaction and loneliness in community-dwelling older women will be evaluated by applying the group-based multimodal exercise training combined with Otago home-based exercise program including strengthening and balance exercises. The original aspect of this study is the presentation of the results to be obtained by combining the effect of group exercise that creates opportunities for social interaction with the structure of the home based Otago exercise program that ensures its sustainability in the home environment.

DETAILED DESCRIPTION:
Within the scope of the program, which will last for 16 weeks, 3 days a week, a total of 48 sessions will be held. The program will be held one day a week with a maximum of 8 participants, under the supervision of a physiotherapist, in the Kadıköy Municipality Social Life House, in the form of group exercise training, and two days a week at the participants' homes, with the implementation of the Otago Home Exercise Program unattended. Participants will be informed that the program should be implemented on non-consecutive days. All warm-up and strengthening exercises will be applied in combination with breathing. While the home exercise program is being taught to the patients, information will be given about the situations where the exercise is contraindicated and should be stopped.

Within the scope of group exercise training, it is planned to implement a structured program of approximately 45-60 minutes, including warm-up, strengthening, balance and cooling exercises.

The control group will not be included in any exercise application, and they will be informed that they can participate in the same program after 16 weeks if they prefer. At the same time, a one-session training will be given to all participants in the application and control groups at the Kadıköy Municipality Social Life House, where information about the factors that increase the risk of falling and house arrangements will be provided.

ELIGIBILITY:
Inclusion Criteria:

* 65 years and older and female gender,
* No cognitive deficit (Montreal Cognitive Assessment (MoCA) score above 21),
* Able to walk without using assistive devices
* those people who can speak and understand Turkish is planned to include in the study.

Exclusion Criteria:

* Patients with unstable cardiovascular disease (unstable angina pectoris, critical aortic stenosis, uncontrolled atrial or ventricular arrhythmia, 3rd degree atrioventricular block, etc.)
* Having a history of fracture in the upper and/or lower extremity up to 1 year ago,
* Neurological, pulmonary, cardiovascular, rheumatological and musculoskeletal diseases that prevent participation in exercise,
* Have a clinical diagnosis that will affect the nervous system, vestibular system or visual balance
* Those with malignancies affecting the lower extremity,
* Those who cannot communicate
* people who participate in physical exercise programs such as pilates, tai-chi, fitness for more than 60 minutes a week is planned not to include in the study.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — Only community-dwelling older women will be recruited in this study.
Enrollment: 76 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-06-17 (Actual)

PRIMARY OUTCOMES:
4-meter Walk Test | Change from initial of the treatment at 16 weeks of treatment
  4 meter Walk Test: The person will be asked to walk the 4-meter distance at his normal speed as in his daily life, and the walking time of the 4-meter distance will be recorded in seconds. This measurement will be utilized to obtain Brief Physical Performance Scale scoring.
5 Times Sit and Stand Test | Change from initial of the treatment at 16 weeks of treatment
  5 times sit and stand test: The patient sits with his arms crossed over his shoulders and his back against a chair. With the "Start" command, the patient is expected to stand up and sit up quickly five times from the standard chair. The elapsed time will be measured with a stopwatch and recorded in seconds.
  This measurement will be utilized to obtain Brief Physical Performance Scale scoring.
One Foot Balance Test | Change from initial of the treatment at 16 weeks of treatment
  Single Leg Balance Test: the participant will be asked to stand on one leg while the knee is in 90° flexion. The stopwatch will be recorded time in seconds. The test will be terminated if the elder's upper foot touches the ground. Separate measurements are made for both extremities.
  This measurement will be utilized to obtain Brief Physical Performance Scale scoring.
Tandem Balance Test | Change from initial of the treatment at 16 weeks of treatment
  Tandem Balance Test: The elder will be asked to stand for 10 seconds with one foot in front of the other. Right leg first and left leg first will be measured separately. This measurement will be utilized to obtain Brief Physical Performance Scale scoring.
Semi-tandem Balance Test | Change from initial of the treatment at 16 weeks of treatment
  Semi-Tandem Balance Test: The elder will be asked to stand for 10 seconds with the heel of one foot beside the other's big toe. Right leg first and the left leg first will be measured separately.
  This measurement will be utilized to obtain Brief Physical Performance Scale scoring.
Timed Get Up and Go Test | Change from initial of the treatment at 16 weeks of treatment
  Timed Get Up and Go Test In the timed get up and go test, a point was marked 3 m from the chair where the participant was sitting. The participant will be asked to get up from the chair and walk 3 m and return to sit on the chair again, and the time to complete the test will be measured with a stopwatch. Times of fourteen seconds or more will be considered as a high risk of falling (Podsiadlo, 1991).

SECONDARY OUTCOMES:
Fear of falling (Activity-Specific Balance Confidence Scale) | Change from initial of the treatment at 16 weeks of treatment
  Activity-Specific Balance Confidence Scale
  Individuals are asked 16 questions about daily living activities inside and outside the home. These activities are; daily activities such as walking around the house, going up and down the stairs, getting on and off the vehicle, climbing uphill, walking in the crowd, walking on the icy pavement, reaching for things at head and eye level in the house. Turkish validity and reliability were established (Karapolat, 2010). For each question, individuals are asked to rate their confidence in the activity between 0 and 100%. These values will be added and divided by 16 and the nearest decimal value will be accepted as the value of the scale. The higher the score, the higher the balance confidence of the individuals.
Hand grip strength (Jamar) | Change from initial of the treatment at 16 weeks of treatment
  The Jamar hand dynamometer, which is recommended by the American Association of Hand Therapists (AETD) and has high validity and reliability in many studies, and therefore accepted as the gold standard, will be used to measure hand grip strength.
  Measurement of hand grip and finger grip strengths, which is the standard position recommended by AETD; in sitting position, shoulder in adduction and neutral rotation, elbow in 90º flexion, forearm in midrotation and supported, and wrist in neutral. In the test procedure, 2 measurements will be made with one minute intervals between each measurement for hand grip and finger grip strengths and the averages will be recorded (Rothstein, 1993).
Quadriceps isometric strength (Microfet) | Change from initial of the treatment at 16 weeks of treatment
  Quadriceps Isometric Strength Assessment
  Microfet 3 hand dynamometer will be used for quadriceps muscle strength. Subjects will be seated in a chair with high armrests, with their knees and hips flexed to 90 degrees. Subjects will be asked to straighten their knees using all their strength, with the hand dynamometer above the ankle. Three separate measurements will be made for the right and left Quadriceps. They will be asked to rest for 10 seconds between each measurement to avoid fatigue. Verbal instructions for each test will be standardized and a loud command will be given: "Push as hard as you can, as hard as you can, as hard as you can" (Deones, 1994).
Fall rating (How many times have you fallen in the last 6 months? Have you been injured after falling?) | Change from initial of the treatment at 16 weeks of treatment
  The number of falling in the past 6 months and fall-related injuries of participants will be questioned.
Participation (World Health Organization Quality of Life Scale Elderly Module-WHOQL-OLD) | Change from initial of the treatment at 16 weeks of treatment
  WHOQL-OLD (Participation) The dimension of "social participation" especially describes being able to participate in daily life activities in society. The WHOQOL-OLD module consists of 24 questions in six dimensions, the answers of which are determined by a five-point Likert scale. These six dimensions are: "sensory functions" (questions 1, 2, 10 and 20), "Autonomy" (questions 3, 4, 5 and 11), "Past, Present, Future Activities" (12, 13, 15) and 19), "Social participation" (questions 14, 16, 17 and 18), "death and dying" (questions 6, 7, 8 and 9) and "Intimacy" (Questions 21, 22, 23 and 24) numbered questions). Possible dimension scores range from 4-20. In addition, the "total score" can be calculated by adding the individual score values. As the score increases, the quality of life also improves (Eser, 2010).
Satisfaction with Life (Satisfaction with Life Scale) | Change from initial of the treatment at 16 weeks of treatment
  Life Satisfaction Scale Diener et al. (1985) and adapted into Turkish by Yetim (1993), the 'Satisfaction with Life Scale' was used. The scale consisting of 5 items; It was prepared in 7-point Likert type and scoring was done accordingly. Likert options "Strongly Disagree (1)", "Disagree (2)", "Partly Disagree (3)", "Undecided (4)", "Partly Agree (5)", "Agree (6)" and "Strongly Agree" It is listed as (7)". The highest score that can be obtained from the scale is 35 (Dağlı, 2016).
Loneliness (UCLA Loneliness Scale- Short Form) | Change from initial of the treatment at 16 weeks of treatment
  UCLA Loneliness Scale- Short Form UCLA-KF is the short form of the scale developed by Russell, Peplau and Cutrona (1980) to determine the general loneliness levels of individuals, and converted into short form by Hays and DiMatteo (1987). The adaptation of the scale to Turkish culture was done by Yıldız and Duy (2014) (Doğan, 2011). UCLA-KF consists of 7 items and should be scored on a 4-point Likert scale. The scoring of the statements in the scale ranges from "Never (1)" to "Always (4)". The lowest score that can be obtained from the scale is 7, and the highest score is 28. An increase in the score obtained from the scale indicates an increase in the level of loneliness.

CONTACTS AND LOCATIONS:
Overall Officials: Nazlı Güngör, PT, MSc, Principal Investigator — Istanbul Arel University
Locations (1):
- Istanbul Arel University, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Buatois S, Perret-Guillaume C, Gueguen R, Miget P, Vancon G, Perrin P, Benetos A. A simple clinical scale to stratify risk of recurrent falls in community-dwelling adults aged 65 years and older. Phys Ther. 2010 Apr;90(4):550-60. doi: 10.2522/ptj.20090158. Epub 2010 Mar 4. PMID 20203094
- [Result] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Result] Cruz-Jimenez M. Normal Changes in Gait and Mobility Problems in the Elderly. Phys Med Rehabil Clin N Am. 2017 Nov;28(4):713-725. doi: 10.1016/j.pmr.2017.06.005. PMID 29031338
- [Result] Deones VL, Wiley SC, Worrell T. Assessment of quadriceps muscle performance by a hand-held dynamometer and an isokinetic dynamometer. J Orthop Sports Phys Ther. 1994 Dec;20(6):296-301. doi: 10.2519/jospt.1994.20.6.296. PMID 7849749
- [Result] Eckstrom E, Neukam S, Kalin L, Wright J. Physical Activity and Healthy Aging. Clin Geriatr Med. 2020 Nov;36(4):671-683. doi: 10.1016/j.cger.2020.06.009. Epub 2020 Aug 19. PMID 33010902
- [Result] Subias-Perie J, Navarrete-Villanueva D, Gomez-Cabello A, Vicente-Rodriguez G, Casajus JA. Health economic evaluation of exercise interventions in people over 60 years old: A systematic review. Exp Gerontol. 2022 May;161:111713. doi: 10.1016/j.exger.2022.111713. Epub 2022 Jan 29. PMID 35104563
- [Result] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356
- [Result] Karapolat H, Eyigor S, Kirazli Y, Celebisoy N, Bilgen C, Kirazli T. Reliability, validity, and sensitivity to change of Turkish Activities-specific Balance Confidence Scale in patients with unilateral peripheral vestibular disease. Int J Rehabil Res. 2010 Mar;33(1):12-8. doi: 10.1097/mrr.0b013e32832c0d72. PMID 20183891
- [Result] Kyrdalen IL, Moen K, Roysland AS, Helbostad JL. The Otago Exercise Program performed as group training versus home training in fall-prone older people: a randomized controlled Trial. Physiother Res Int. 2014 Jun;19(2):108-16. doi: 10.1002/pri.1571. Epub 2013 Dec 11. PMID 24339273
- [Result] Kocic M, Stojanovic Z, Nikolic D, Lazovic M, Grbic R, Dimitrijevic L, Milenkovic M. The effectiveness of group Otago exercise program on physical function in nursing home residents older than 65years: A randomized controlled trial. Arch Gerontol Geriatr. 2018 Mar-Apr;75:112-118. doi: 10.1016/j.archger.2017.12.001. Epub 2017 Dec 10. PMID 29241091
- [Result] Latham NK, Bennett DA, Stretton CM, Anderson CS. Systematic review of progressive resistance strength training in older adults. J Gerontol A Biol Sci Med Sci. 2004 Jan;59(1):48-61. doi: 10.1093/gerona/59.1.m48. PMID 14718486
- [Result] Lord SR, Delbaere K, Sturnieks DL. Aging. Handb Clin Neurol. 2018;159:157-171. doi: 10.1016/B978-0-444-63916-5.00010-0. PMID 30482312
- [Result] Makanae Y, Fujita S. Role of Exercise and Nutrition in the Prevention of Sarcopenia. J Nutr Sci Vitaminol (Tokyo). 2015;61 Suppl:S125-7. doi: 10.3177/jnsv.61.S125. PMID 26598823
- [Result] Michikawa T, Nishiwaki Y, Takebayashi T, Toyama Y. One-leg standing test for elderly populations. J Orthop Sci. 2009 Sep;14(5):675-85. doi: 10.1007/s00776-009-1371-6. Epub 2009 Oct 3. PMID 19802686
- [Result] Papa EV, Dong X, Hassan M. Resistance training for activity limitations in older adults with skeletal muscle function deficits: a systematic review. Clin Interv Aging. 2017 Jun 13;12:955-961. doi: 10.2147/CIA.S104674. eCollection 2017. PMID 28670114
- [Result] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Result] Rodrigues F, Domingos C, Monteiro D, Morouco P. A Review on Aging, Sarcopenia, Falls, and Resistance Training in Community-Dwelling Older Adults. Int J Environ Res Public Health. 2022 Jan 13;19(2):874. doi: 10.3390/ijerph19020874. PMID 35055695
- [Result] Shubert TE. Evidence-based exercise prescription for balance and falls prevention: a current review of the literature. J Geriatr Phys Ther. 2011 Jul-Sep;34(3):100-8. doi: 10.1519/JPT.0b013e31822938ac. PMID 22267151
- [Result] Thomas S, Mackintosh S, Halbert J. Does the 'Otago exercise programme' reduce mortality and falls in older adults?: a systematic review and meta-analysis. Age Ageing. 2010 Nov;39(6):681-7. doi: 10.1093/ageing/afq102. Epub 2010 Sep 4. PMID 20817938
- [Result] Unver B, Baris RH, Yuksel E, Cekmece S, Kalkan S, Karatosun V. Reliability of 4-meter and 10-meter walk tests after lower extremity surgery. Disabil Rehabil. 2017 Dec;39(25):2572-2576. doi: 10.1080/09638288.2016.1236153. Epub 2016 Oct 11. PMID 27728985
- [Result] Yang Y, Wang K, Liu H, Qu J, Wang Y, Chen P, Zhang T, Luo J. The impact of Otago exercise programme on the prevention of falls in older adult: A systematic review. Front Public Health. 2022 Oct 20;10:953593. doi: 10.3389/fpubh.2022.953593. eCollection 2022. PMID 36339194